CLINICAL TRIAL: NCT05787041
Title: The Effect of High Fat Diet on the Pharmacokinetics of AD16 Tablets in Healthy Chinese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: South China Center For Innovative Pharmaceuticals (Other)
Collaborators: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCCIP-AD16-2018-02
Record Dates: First submitted 2023-03-01; First posted 2023-03-28 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fat diet group (Experimental): A single dose of AD16 tablets was taken orally after a high fat diet
  Interventions: Other: high-fat diet group（AD16 20mg）
- Fasting group (Experimental): A single dose of AD16 tablets was taken orally under fasting conditions
  Interventions: Other: fasted group（AD16 20mg）

INTERVENTIONS:
Other: high-fat diet group（AD16 20mg） — AD16 was administered with 240 mL water 30 minutes after the subjects ate a high-fat, high-calorie food.
  Arms: High-fat diet group
Other: fasted group（AD16 20mg） — Subjects took AD16 on an empty stomach and fasted within 4 hours after taking the drug.
  Arms: Fasting group

SUMMARY:
The study was a single-center, randomized, open-access, two-crossover, single-dose study design with 16 subjects to evaluate the pharmacokinetics of a high-fat diet on a single dose of oral AD16 tablets in healthy Chinese adults and the safety of a single dose of oral AD16 tablets in healthy Chinese adults.

Compared with fasting administration, a high-fat diet reduced the rate of AD16 tablet absorption in healthy adult subjects and had no effect on overall exposure to AD16.

The elimination and distribution characteristics of AD16 in vivo were similar under the conditions of feeding and fasting administration.

A single dose of AD16 tablets after fasting and high fat diet showed good safety.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Healthy subjects were aged 18-45 years (including boundary values), male and female.
2. Weight ≥50kg (male) or ≥45kg (female), and body mass index (BMI) of 19-24kg/m2 (including the boundary values at both ends).
3. Have fully understood this study, voluntarily participated in it, and signed the Informed Consent.
4. Subjects are able to communicate well with researchers and complete the study according to protocol.
5. The subjects were deemed to be in good health based on physical examination, medical history, vital signs, electrocardiogram, chest X-ray, abdominal ultrasound, and laboratory tests.
6. Subject (including partner) is willing to have no pregnancy plan for the next 30 days (female subject) or 90 days (male subject) and is willing to use effective contraception.

Exclusion Criteria:

1. Positive for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody or HIV antibody.
2. The patient has symptoms or related history of any serious disease, including but not limited to heart, liver, kidney, or other acute or chronic digestive tract or respiratory tract diseases, as well as diseases of the blood, endocrine, neurological, psychiatric and other systems, or any other disease or physiological condition that can interfere with the study results.
3. A history of postural hypotension with frequent episodes.
4. A history of frequent nausea or vomiting due to any cause.
5. Any clear history of drug or food allergies, especially allergies to ingredients similar to the drugs in this study.
6. Have special dietary requirements and cannot comply with the uniform diet provided by the clinical research center.
7. Previous drug abuse history or positive urine drug screening during screening period.
8. Smokers who smoked more than 5 cigarettes a day in the 3 months before the test.
9. Heavy drinkers or regular drinkers in the 6 months prior to the study screening, who drank more than 14 units of alcohol per week (1 unit of alcohol ≈360 mL beer or 45 mL 40% spirits or 150 mL wine) or had a positive alcohol breath test during the screening period.
10. Excessive consumption of tea, coffee (more than 6 cups) and/or caffeinated beverages (more than 1L) per day.
11. Take food or drink rich in xanthine, grapefruit or alcohol, caffeine (e.g., dragon fruit, mango, grapefruit, chocolate, coffee or tea) within 48 hours before administration.
12. Surgical procedures, transfusions of blood or blood components in the month prior to study screening.
13. Blood loss or donation of more than 400 mL in the 2 months prior to screening.
14. Participated in other clinical studies and took experimental drugs within 3 months prior to study screening.
15. Study participants who had received any medication in the 28 days prior to screening.
16. Pregnant or lactating women or women who have had unprotected sex within 14 days.
17. Those unable to complete the study for other reasons or deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Cmax of AD16 | Up to Day 10
  Maximum (peak) plasma drug concentration
AUC 0-t of AD16 | Up to Day 10
  Area under the plasma concentration-time curve(AUC) from time zero to time t
AUC 0-∞ of AD16 | Up to Day 10
  Area under the plasma concentration-time curve(AUC) from time zero to infinity
t1/2 of AD16 | Up to Day 10
  Elimination half-life (to be used in a one-compartment or noncompartmental model)
Tmax of AD16 | Up to Day 10
  Time to reach the maximum (peak) plasma concentration following drug administration
CL/F of AD16 | Up to Day 10
  CL/F is defined as the ratio of total clearance(CL) to bioavailability(F).
Vd/F of AD16 | Up to Day 10
  Apparent volume of distribution after non-intravenous administration
MRT of AD16 | Up to Day 10
  Mean residence time(MRT)
λz of AD16 | Up to Day 10
  Terminal disposition rate constant/terminal rate constant

SECONDARY OUTCOMES:
Adverse events | day-7 to day 10
  The number of adverse events
Serious adverse events | day-7 to day 10
  The number of serious adverse events
Number of participants with abnormal laboratory test results | day-7 to day-1 and day10
  Laboratory tests include blood routine, blood biochemistry, coagulation function and urine routine
Number of participants with abnormal vital signs | day-7 to day3 and day7 to day10
  vital signs include Pulse, blood pressure, body temperature and respiratory rate were observed at different time points before and after medication.
Number of participants with abnormal 12- Lead ECG readings | day-7 to day-1 and days3 、10
  abnormal 12- Lead ECG
Number of participants with abnormal physical examination findings | day-7 to day-1 and day10
  The skin, mucosa, lymph nodes, head, neck, chest, abdomen, spine/limbs and nervous system were observed at different time points before and after medication.
Concomitant medication | Up to Day 10
  Any concomitant medication

CONTACTS AND LOCATIONS:
Locations (1):
- The Central South University Xiang Ya Hospital, Changsha, China

REFERENCES:
- [Derived] Peng D, Xu S, Zou T, Wang Y, Ouyang W, Zhang Y, Dong C, Li D, Guo J, Shen Q, Hu X, Zhou W, Li X, Qin Q. Safety, tolerability, pharmacokinetics and effects of diet on AD16, a novel neuroinflammatory inhibitor for Alzheimer's disease: a randomized phase 1 study. BMC Med. 2023 Nov 23;21(1):459. doi: 10.1186/s12916-023-03126-9. PMID 37996817